CLINICAL TRIAL: NCT05802342
Title: a Multicenter, Randomized, Double-blind Phase II Trial To Evaluate Monosialate Tetrahexose-ganglioside Sodium Injection (GM1) for Prevention of Peripheral Neuropathy in Patients With Breast Cancer Induced by Albumin-bound Paclitaxel Regimen Adjuvant/Neoadjuvant Therapy
Brief Title: A Multicenter, Randomized, Double-blind Phase II Trial to Evaluate GM1 Prevention of Peripheral Neuropathy in Patients With Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GM1-CIPN-202
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: To Evaluate the Effectiveness of GM1 in the Prevention of Albumin-paclitaxel Therapy Induced Peripheral Neuropathy in Breast Cancer Patients

STUDY DESIGN:
Intervention Model Description: This study was randomly divided into 3 groups at 1:1:1 with 50 subjects in each group. The treatment plan was as follows.
  Group A: GM1 (100 mg) + albumin paclitaxel; Group B: GM1 (400 mg) + albumin paclitaxel; Group C: placebo + albumin paclitaxel;
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): GM1 (100 mg) + albumin paclitaxel
  Interventions: Drug: Monosialotetrahexose ganglioside sodium injection
- B (Experimental): GM1 (400 mg) + albumin paclitaxel
  Interventions: Drug: Monosialotetrahexose ganglioside sodium injection
- C (Placebo Comparator): placebo + albumin paclitaxel
  Interventions: Drug: Monosialotetrahexose ganglioside sodium injection

INTERVENTIONS:
Drug: Monosialotetrahexose ganglioside sodium injection — The treatment period was GM1/ placebo with albumin-paclitaxel from cycle 1 to cycle 4/6. The treatment period was GM1/ placebo with albumin-paclitaxel. GM1/ placebo was administered every 2 weeks /3 weeks. GM1 / placebo was administered 1 day before administration (D0), on the day of administration (D1) and on the day after administration (D2), and albumin-paclitaxel-based chemotherapy was administered from day 1, with a total of 4/6 cycles of administration. GM1/ placebo was administered every 2 weeks /3 weeks. GM1 / placebo was administered 1 day before administration (D0), on the day of administration (D1) and on the day after administration (D2), and albumin-paclitaxel-based chemotherapy was administered from day 1, with a total of 4/6 cycles of administration.

SUMMARY:
This randomized, double-blind, multicenter, placebo-controlled Phase II trial was designed to investigate the efficacy and safety of GM1 in the prevention of peripheral neuropathy caused by albumin-bound paclitaxel regimen in breast cancer patients.This study was randomly divided into 3 groups at 1:1:1 with 50 subjects in each group Subjects received study treatment until the end of treatment for a total of 4/6 cycles. The treatment period was GM1/ placebo combined with albumin-bound paclitaxel therapy. GM1 / placebo was administered 1 day before administration (D0), on the day of administration (D1) and on the day after administration (D2), and albumin-bound paclitaxel was administered starting on day D1, with a total of 4/6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the content of the experiment and voluntarily sign the informed consent;
2. Age from 18 to 75 years old (including both ends);
3. Breast cancer patients who provide definitive histological and/or cytological diagnosis of breast cancer and are proposing adjuvant/neoadjuvant therapy with the albumin-paclitaxel regimen;
4. ECOG score 0~1;
5. The organ function level must meet the requirements
6. Subjects (both male and female) agreed to use effective contraception from the time of signing the informed consent to 30 days after the last use of the study drug. Female subjects of childbearing age cannot be pregnant or lactating.
7. Patients can accurately record or express the occurrence and severity of neurotoxicity in questionnaires;
8. After enrollment, patients should not receive other treatments or care that might prevent or treat neurotoxic adverse events

Exclusion Criteria:

1. Presence of grade 1 peripheral neurotoxicity (CTCAE≥1) or symptoms of peripheral neuropathy (FACT/GOG-Ntx≥1)
2. There are risk factors for peripheral neuropathy (except peripheral neuropathy caused by chemotherapy),Including but not limited to: diabetic peripheral neuropathy; Peripheral vascular disease; Folic acid, B12 vitamin deficiency; Postoperative neuropathy; Post-traumatic neuropathy; Peripheral neuroinflammatory lesions; Peripheral neuropathy caused by tumor compression and infiltration; Other researchers believe that can cause limb pain, numbness, paresthesia, dysfunction of the skin, muscle, vascular diseases;
3. Cardiovascular and cerebrovascular diseases, including but not limited to: Myocardial infarction (within 6 months before signing the informed consent), unstable angina, high risk of uncontrollable arrhythmia, coronary artery bypass grafting, cerebrovascular accident (within 6 months before signing the informed consent), congestive heart failure (cardiac function grade III-Ⅳ), pulmonary embolism, deep vein thrombosis, and other cardiovascular and cerebrovascular systems deemed unsuitable for inclusion by the investigator General disease;
4. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) after optimal treatment with antihypertensive drugs; Patients with blood pressure deemed unsuitable for clinical trials by the investigator;
5. Diabetic patients with HBA1c ≥9.0%;
6. Active bacterial, fungal, or viral infections that require systematic treatment within one week prior to initial administration; Infectious diarrhea occurred within 4 weeks prior to initial administration;
7. History of inherited abnormal glucose and lipid metabolism (ganglioside accumulation disease, such as familial amaurosis, retinal degeneration) or autoimmune disease;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); Syphilis antibody positive;
9. Active hepatitis B (HBsAg positive with HBV-DNA > 500 IU/ml or lower limit of Center detection [only when lower limit of Center detection is higher than 500 IU/ml]), active hepatitis C (patients with HCV antibody positive but HCV-RNA < lower limit of Center detection are admitted);
10. Known allergy to ganglioside drugs or any excipient component of such products; Or to treat an allergy to a drug or any excipient component of such product;
11. Patients who, in the judgment of the investigator, may increase the risk associated with the study, may interfere with the interpretation of the study results, or may be deemed unsuitable for inclusion by the investigator and/or sponsor.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Grade ≥2 neurotoxicity （CTCAE） | C4D3
The difference between the FACT/GOG-Ntx score and the baseline score | C4D3

SECONDARY OUTCOMES:
The incidence of peripheral neurotoxicity during cycles 1 to 6 and follow-up | 12 month
Change in FACT/GOG-Ntx scores from baseline during 1-6 cycles and follow-up | 12 month
Change in CIPN20 score from baseline after 1-6 cycles and follow-up | 12 month
incidence of adverse events | 12 month

IPD SHARING:
Plan to Share IPD: No